CLINICAL TRIAL: NCT03103724
Title: A Phase II Study Evaluating the Efficacy of Enzalutamide and the Role of ARv7 in Metastatic Castration Resistant Prostate Cancer (mCRPC) Patients With Visceral Disease.
Acronym: EXCALIBUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 178-15
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enzalutamide (Experimental): All subjects will receive open label enzalutamide 160 mg (4 x 40 mg capsules), orally once daily.
  Interventions: Drug: Xtandi

INTERVENTIONS:
Drug: Xtandi — Enzalutamide 160 mg (4 x 40 mg capsules), orally once daily
  Other Names: Enzalutamide

SUMMARY:
Open label, single arm, phase II multicentre study designed to determine the clinical benefit, as measured by 3-months disease control rate (DCR) provided by enzalutamide in metastatic Castration Resistant Prostate Cancer patients with at least one visceral site involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. ECOG PS 0-1-2
3. Biopsy (primary tumour or metastases) confirming the diagnosis of prostate adenocarcinoma
4. Documented measurable metastatic visceral disease (according to RECIST 1.1 criteria) considering metastases in lung or liver or extraregional lymphnodes
5. Written informed consent
6. Platelets > or = 100 x109/L; haemoglobin > or = 9 g/dl; neutrophils > or 1.5 x 109/L
7. Bilirubin < or = 2 mg/dl, AST and ALT < or = 2.5 times the UNL or < or = 5 times UNL for pts with liver metastases; serum albumin > or = the LNL
8. Patients of childbearing age should use contraceptive methods
9. Life expectancy > 3 months
10. Able to swallow the study drug and comply with study requirements;
11. Willing and able to give informed consent.
12. Ongoing androgen deprivation therapy with a GnRH analogue or orchiectomy (i.e., surgical or medical castration);
13. Patients may have received previous therapy including chemotherapy (docetaxel) last cycle must be received 3 weeks before start of experimental treatment. Hormonal treatment containing bicalutamide must be interrupted 2 weeks before start of study therapy
14. Previous radiotherapy (prostate and/or bone) is accepted but must be interrupted 3 weeks before start of experimental treatment.
15. Serum testosterone level < 1.7 nmol/L (50 ng/dL) at the Screening visit
16. Progressive disease by PSA or imaging in the setting of medical or surgical castration. Disease progression for study entry is defined as one or more of the following three criteria (according with PCWG2):

    * PSA progression defined by a minimum of three rising PSA levels with an interval of ≥ 1 week between each determination. The PSA value at the Screening visit should be ≥ 2 g/L (2 ng/ml); if the third PSA value is less than second PSA, a fourth PSA must be repeated and if it the value is higher than second must be considered as disease
    * Soft tissue/visceral disease progression defined by RECIST 1.1;
    * Bone disease progression defined by two or more new lesions on bone scan.

Exclusion Criteria:

1. Severe, concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment;
2. Metastases in the brain or active epidural disease;
3. History of another malignancy within the previous 5 years other than curatively treated non-melanomatous skin cancer;
4. History of seizure, including any febrile seizure, loss of consciousness, or transient ischemia attack within 12 months of enrollment (Day 1 visit), or any condition that may pre-dispose to seizure (e.g., prior stroke, head trauma with loss of consciousness requiring hospitalization);
5. Clinically significant cardiovascular disease including: Myocardial infarction within 6 months; Uncontrolled angina within 3 months; Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within 3 months results in a left ventricular ejection fraction that is ≥ 45%;
6. Diagnosed or suspected congenital long QT syndrome;
7. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
8. Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer within last 3 months);
9. Major surgery within 4 weeks prior to enrollment (Day 1 visit);
10. Prior treatment with abiraterone acetate;
11. Participation in a clinical trial about an experimental anti-androgen agent (eg. ARN-509, ODM-201, VT-464, except for placebo arm);
12. Treatment (concomitant or in the previous 2 weeks) with anti-androgens (eg. Bicalutamide, nilutamide, flutamide) or 5-a reductase inhibitors (eg. finasteride, dutasteride).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 3 months
  To determine the clinical benefit, as measured by 3 months disease control rate (DCR) provided by enzalutamide in mCRPC patients with visceral disease.

SECONDARY OUTCOMES:
Safety of the treatment per NCI-CTCA v. 4.0 | 2 years
  To determine the safety of the treatment according to NCI-CTCA v. 4.0
Quality of life by EQ-5D-5L e FACT-P | 2 years
  To evaluate quality of life as assessed by EQ-5D-5L e FACT-P questionnaire
Pain assessment | 2 years
  To evaluate pain as assessed by BPI-SF questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elena Verzoni, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori Milano
Locations (1):
- Elena Verzoni, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Astellas Pharma Ltd. Xtandi (enzalutamide) 40mg soft capsules. Summary of Product Characteristics. 26 June 2013.
- [Result] Ahmed M, Li LC. Adaptation and clonal selection models of castration-resistant prostate cancer: current perspective. Int J Urol. 2013 Apr;20(4):362-71. doi: 10.1111/iju.12005. Epub 2012 Nov 19. PMID 23163774
- [Result] Antonarakis ES, Lu C, Wang H, Luber B, Nakazawa M, Roeser JC, Chen Y, Mohammad TA, Chen Y, Fedor HL, Lotan TL, Zheng Q, De Marzo AM, Isaacs JT, Isaacs WB, Nadal R, Paller CJ, Denmeade SR, Carducci MA, Eisenberger MA, Luo J. AR-V7 and resistance to enzalutamide and abiraterone in prostate cancer. N Engl J Med. 2014 Sep 11;371(11):1028-38. doi: 10.1056/NEJMoa1315815. Epub 2014 Sep 3. PMID 25184630
- [Result] Arlen PM, Bianco F, Dahut WL, D'Amico A, Figg WD, Freedland SJ, Gulley JL, Kantoff PW, Kattan MW, Lee A, Regan MM, Sartor O; Prostate Specific Antigen Working Group. Prostate Specific Antigen Working Group guidelines on prostate specific antigen doubling time. J Urol. 2008 Jun;179(6):2181-5; discussion 2185-6. doi: 10.1016/j.juro.2008.01.099. Epub 2008 Apr 18. PMID 18423743
- [Result] Beer TM, Tombal B. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Oct 30;371(18):1755-6. doi: 10.1056/NEJMc1410239. No abstract available. PMID 25354111
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Ferlay J, Parkin DM, Steliarova-Foucher E. Estimates of cancer incidence and mortality in Europe in 2008. Eur J Cancer. 2010 Mar;46(4):765-81. doi: 10.1016/j.ejca.2009.12.014. Epub 2010 Jan 29. PMID 20116997
- [Result] Fitzpatrick JM, de Wit R. Taxane mechanisms of action: potential implications for treatment sequencing in metastatic castration-resistant prostate cancer. Eur Urol. 2014 Jun;65(6):1198-204. doi: 10.1016/j.eururo.2013.07.022. Epub 2013 Jul 25. PMID 23910941
- [Result] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. Part II: Treatment of advanced, relapsing, and castration-resistant prostate cancer. Eur Urol. 2014 Feb;65(2):467-79. doi: 10.1016/j.eururo.2013.11.002. Epub 2013 Nov 12. PMID 24321502
- [Result] Horwich A, Parker C, de Reijke T, Kataja V; ESMO Guidelines Working Group. Prostate cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi106-14. doi: 10.1093/annonc/mdt208. Epub 2013 Jun 27. No abstract available. PMID 23813930
- [Result] Huggins C, Hodges CV. Studies on prostatic cancer. I. The effect of castration, of estrogen and of androgen injection on serum phosphatases in metastatic carcinoma of the prostate. 1941. J Urol. 2002 Feb;167(2 Pt 2):948-51; discussion 952. No abstract available. PMID 11905923
- [Result] Kuczynski EA, Sargent DJ, Grothey A, Kerbel RS. Drug rechallenge and treatment beyond progression--implications for drug resistance. Nat Rev Clin Oncol. 2013 Oct;10(10):571-87. doi: 10.1038/nrclinonc.2013.158. Epub 2013 Sep 3. PMID 23999218
- [Result] Merseburger AS, Bellmunt J, Jenkins C, Parker C, Fitzpatrick JM; European Treatment Practices Group. Perspectives on treatment of metastatic castration-resistant prostate cancer. Oncologist. 2013;18(5):558-67. doi: 10.1634/theoncologist.2012-0478. Epub 2013 May 13. PMID 23671006
- [Result] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Result] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Result] Ryan CJ, Tindall DJ. Androgen receptor rediscovered: the new biology and targeting the androgen receptor therapeutically. J Clin Oncol. 2011 Sep 20;29(27):3651-8. doi: 10.1200/JCO.2011.35.2005. Epub 2011 Aug 22. PMID 21859989
- [Result] Scher HI, Beer TM, Higano CS, Anand A, Taplin ME, Efstathiou E, Rathkopf D, Shelkey J, Yu EY, Alumkal J, Hung D, Hirmand M, Seely L, Morris MJ, Danila DC, Humm J, Larson S, Fleisher M, Sawyers CL; Prostate Cancer Foundation/Department of Defense Prostate Cancer Clinical Trials Consortium. Antitumour activity of MDV3100 in castration-resistant prostate cancer: a phase 1-2 study. Lancet. 2010 Apr 24;375(9724):1437-46. doi: 10.1016/S0140-6736(10)60172-9. Epub 2010 Apr 14. PMID 20398925
- [Result] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Derived] Sepe P, Procopio G, Pircher CC, Basso U, Caffo O, Cappelletti V, Claps M, De Giorgi U, Fratino L, Guadalupi V, Miodini P, De Marco C, Perrucci B, Mennitto A, Santini D, Spina F, Stellato M, de Braud F, Verzoni E. A phase II study evaluating the efficacy of enzalutamide and the role of liquid biopsy for evaluation of ARv7 in mCRPC patients with measurable metastases including visceral disease (Excalibur study). Ther Adv Med Oncol. 2024 Jan 22;16:17588359231217958. doi: 10.1177/17588359231217958. eCollection 2024. PMID 38264520